CLINICAL TRIAL: NCT04319848
Title: Safety and Efficacy of Tissue Engineered Endothelial Keratoplasty (TE-EK)
Brief Title: Safety and Efficacy of Tissue Engineered Endothelial Keratoplasty
Acronym: TE-EK
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Jodhbir Mehta, Senior Consultant Head Corneal and External Eye Disease and Refractive Service, Singapore Eye Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1391/77/2016
Record Dates: First submitted 2017-11-19; First posted 2020-03-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Mild to Moderate Corneal Endothelial Decompensation; Bullous Keratopathy; Fuchs' Endothelial Dystrophy; Post-surgical Corneal Decompensation (Irreversible)
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Intervention Model Description: interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TE-EK treatment group (Experimental): The TE-EK surgery will be performed by the Principle Investigator with a standard DSAEK technique. The PI has performed over 300, EK surgeries and we have previously shown that the corneal endothelial loss rates from the PI are 16% at 1 year with a primary graft failure rates of <1.5%. A patient's participation in the study or not will not change the treatment strategy in any manner.
  Interventions: Other: TE-EK treatment group

INTERVENTIONS:
Other: TE-EK treatment group — Transplantation of tissue-engineered endothelial graft through DSAEK procedure.

SUMMARY:
Assessment of safety and efficacy of tissue-engineered corneal endothelial graft material generated using cultured human corneal endothelial cells for tissue-engineered endothelial keratoplasty (TE-EK).

DETAILED DESCRIPTION:
The specific aim of this clinical trial is to assess the clinical efficacy and safety outcomes of patients receiving Tissue-Engineered Endothelial keratoplasty (TE-EK) graft material generated from human corneal endothelial cells (HCEnCs) propagated in a regulatory-approved dual media approach. Post-operative follow-ups and visits will follow current EK protocols of Singapore National Eye Centre. Clinical assessments include postoperative visual acuity, intraocular pressure, keratometric astigmatism, spherical equivalent, endothelial cell density, anterior segment optical coherence tomography (ASOCT), contrast sensitivity, as well as any postoperative complications such as graft dislocation or primary graft failure.

ELIGIBILITY:
Inclusion Criteria:

Patients who have mild to moderate corneal endothelial decompensation or bullous keratopathy, but with minimal corneal stromal scarring resulting from a variety of conditions including:

* Fuchs' endothelial dystrophy
* Post-surgical corneal decompensation (irreversible) - all forms of pseudophakic or aphakic bullous keratopathy

Exclusion Criteria:

* Severe forms or late stage presentation of corneal decompensation with severe corneal stromal scarring, unsuitable for TE-EK surgery as opposed to penetrating keratoplasty
* Patients with complex anterior segment complications precluding a successful TE-EK procedure
* Patients who have other forms of endothelial dystrophy, traumatic corneal decompensation, or post-inflammatory corneal decompensation
* Post-laser iridotomy or glaucoma related corneal decompensation
* Patients not keen to participate in the clinical trial
* Patients who are below 21 years of age or above 80 years of age
* Patients who are pregnant
* Patients who are cognitively impaired
* Patients who are prisoners
* Patients who are allergic to antibiotics

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
(BSCVA) | 3 months
  BSCVA will be converted to logarithm of the minimum angle of resolution (logMAR) visual acuity for statistical analysis.

SECONDARY OUTCOMES:
Keratometric astigmatism and spherical equivalent | 3 months
  Measured by an autokeratorefractometer (RK-8100; Topcon, Tokyo, Japan)
Intraocular pressure measurement | 3 Months
  Measured by a noncontact tonometry (CT-60; Topcon)
Endothelial cell density (ECD) | 3 months
  Measured by a noncontact specular microscope (Konan Medical Corp, Hyogo, Japan). The ECD data will be expressed as percentage of cell loss compared with the donor ECD.
Graft thickness | 1 month
  Measured by ASOCT (Visante OCT, Carl Zeiss Meditec)
Contrast sensitivity | 6 months
  Pentacam scatter
Postoperative complications | 1 month
  Postoperative complications, such as graft dislocation, graft rejection, will be evaluated with slit lamp biomicroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jodhbir Mehta, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soh YQ, Poh SSJ, Peh GSL, Mehta JS. New Therapies for Corneal Endothelial Diseases: 2020 and Beyond. Cornea. 2021 Nov 1;40(11):1365-1373. doi: 10.1097/ICO.0000000000002687. PMID 34633355